CLINICAL TRIAL: NCT01326767
Title: An Open-Label, Randomized, Parallel Group Study of Patients Treated With Paclitaxel With Standard Dosing Versus Pharmacokinetic Guided Dose Adjustment in Patients With Advanced Non Small Cell Lung Cancer (NSCLC)
Brief Title: Central European Society for Anticancer Research (CESAR) Study of Paclitaxel Therapeutic Drug Monitoring
Acronym: CEPAC-TDM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Central European Society for Anticancer Drug Research (Other)
Collaborators: Saladax Biomedical, Inc. (Industry); Cantonal Hospital of St. Gallen (Other); University Hospital, Basel, Switzerland (Other); Assign Data Management and Biostatistics GmbH (Other); Wake Forest University (Other); University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-III-002; 2010-023688-16 (EudraCT Number)
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel dosing according to SmPC (Active Comparator)
  Interventions: Drug: Paclitaxel dosing according to SmPC
- Individualized pharmacokinetically driven paclitaxel dosing (Experimental): In the first treatment cycle, the Paclitaxel dose is adapted depending on the age and the gender of the patient. In the treatment cycles 2-6 the Paclitaxel dose is adapted based on individual PK data and toxicities.
  Interventions: Drug: Individualized pharmacokinetically driven paclitaxel dosing

INTERVENTIONS:
Drug: Paclitaxel dosing according to SmPC — Paclitaxel i.V. Up to 6 cycles Dosing according to SmPC
  Arms: Paclitaxel dosing according to SmPC
Drug: Individualized pharmacokinetically driven paclitaxel dosing — Paclitaxel i.V. Up to 6 cycles Dosing based on patient age, gender, severity of neutropenia and Paclitaxel plasma concentration
  Arms: Individualized pharmacokinetically driven paclitaxel dosing

SUMMARY:
This study will be performed on grade IIIb and grade IV Non Small Cell Lung Cancer (NSCLC) chemotherapy naive patients with good performance status. In course of this study, patients will be treated with Paclitaxel in combination with either Cisplatin or Carboplatin in a maximum of six therapy cycles. The goal of this study is to determine, if a pharmakokinetic driven dose adaptation of paclitaxel leads to a reduction of of grade 4 neutropenia, compared to conventional Paclitaxel dosing, without affecting progression free survival and overall survival.

This study includes a biomarker analysis and an optional genetic substudy.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the protocol requirements and risks, and providing written informed consent.
* Patients with histologically confirmed NSCLC (stage IIIB-IV).
* Patients considered for first-line palliative chemotherapy with paclitaxel in combination with either cisplatin or carboplatin. Patients having received prior adjuvant non taxane-containing adjuvant chemotherapy are eligible.
* At least one bidimensionally measurable lesion according to RECIST 1.1.
* ECOG Performance Status (ECOG-PS) status ≤ 2.
* Female or male patients of 18 to 75 years of age at randomization
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum pregnancy test within 1 week prior to beginning treatment on this trial. Nursing patients are excluded. Sexually active men must also use acceptable contraceptive methods (condom).
* An absolute neutrophil count >1,500 cells/ mm3 (= 1.5 G/l).
* Platelet count > 100,000/mm3.
* Total bilirubin ≤ 2 x upper limit of normal.
* AST and ALT ≤ 2.5 x upper limit of normal, or ≤ 5 x upper limit of normal in case of liver metastases.
* Creatinine clearance (according to the Cockcroft-Gault formula) ≥30ml/min. For patients planned to receive Cisplatin: Creatinine clearance ≥60ml/min.
* Patients suffering from asymptomatic brain metastases can be enrolled in case corticosteroid therapy is not indicated. Prior irradiation must be completed at least 4 weeks prior to first cycle of treatment.

Exclusion Criteria:

* Serious concomitant systemic disorders (e.g., active infection, severe heart disease, uncontrolled hypertension or diabetes mellitus) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
* A history of hypersensitivity reactions to drugs formulated in polyoxyethylated castor oil.
* Having received prior treatment with paclitaxel or cisplatin or carboplatin (other drugs/drug combinations are allowed).
* Concomitant treatment with any targeted drug (licensed or experimental) like bevacizumab or cetuximab.
* Any condition / concomitant disease not allowing chemotherapy with paclitaxel, the platinum compound (carboplatin or cisplatin) or required premedication for the treatment regimen.
* Pregnant/nursing women.
* Individuals known to be seropositive for human immunodeficiency virus, hepatitis C virus, hepatitis B surface antigen or syphilis.
* Treatment with cytotoxic or biologic agents or any experimental drug within the 4 weeks prior to beginning treatment on this study.
* Secondary malignancy within the last five years, with the exception of adequately treated carcinoma-in-situ of the uterine cervix, basal-cell carcinoma of the skin and pTa or pTis urothelial cancer.
* Medical or psychological conditions that would not permit the patient to complete the study or sign informed consent.
* Preexisting neuropathy > grade I NCI-CTC.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Grad 4 Neutropenia | up to 6 weeks on treatment
  The rate of grade 4 Neutropenia during the second treatment cycle between the conventional Paclitaxel dosing arm and pharmacokinetically driven Paclitaxel dosing arm is compared. At the same time progression free survival and overall survival must not be affected.

SECONDARY OUTCOMES:
Objective tumor response according to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST v1.1) | 24 months
Progression free survival | 24 month
Overall survival | 24 month
Overall neutropenia | 24 month
  Overall neutropenia ( i.e. during total chemotherapy duration) assessed from clinical hematology data and by model-based estimations of individual neutrophil curves
Hematological / non-hematological toxicites | 24 months
  Hematological (leucocytopenia, anemia, thrombocytopenia) and non-hematological toxicities (e.g. neurological, musculosceletal and gastrointestinal adverse events)
Cumulative dose and dose intensity of paclitaxel and platinum drug | 24 months
Incidence of changes from cisplatin to carboplatin and reasons thereof | 24 months
Overall rate of febrile neutropenia and hospitalization due to chemotherapy-associated adverse events | 24 months
Health economic analysis using QoL Questionnaires | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Joerger, MD PhD, Study Chair — Central European Society for Anticancer Drug Research; Ulrich Jaehde, PhD, Study Director — Central European Society for Anticancer Drug Research; Frank Mayer, MD, Principal Investigator — Eberhard-Karls-Universität Tübingen
Locations (11):
- Germany (10):
  - CESAR Study Center, Bochum
  - CESAR study center, Bonn
  - CESAR Study Center, Essen
  - CESAR study center, Gerlingen
  - CESAR study center, Großhansdorf
  - CESAR Study Center, Halle
  - CESAR Study Center, Leer
  - CESAR Study Center, Löwenstein
  - CESAR Study Center, Munich
  - CESAR Study Center, Tübingen
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Derived] Joerger M, von Pawel J, Kraff S, Fischer JR, Eberhardt W, Gauler TC, Mueller L, Reinmuth N, Reck M, Kimmich M, Mayer F, Kopp HG, Behringer DM, Ko YD, Hilger RA, Roessler M, Kloft C, Henrich A, Moritz B, Miller MC, Salamone SJ, Jaehde U. Open-label, randomized study of individualized, pharmacokinetically (PK)-guided dosing of paclitaxel combined with carboplatin or cisplatin in patients with advanced non-small-cell lung cancer (NSCLC). Ann Oncol. 2016 Oct;27(10):1895-902. doi: 10.1093/annonc/mdw290. Epub 2016 Aug 8. PMID 27502710
- See also: CESAR - Homepage — http://www.cesar.or.at/main.asp?VID=1&kat1=11&kat2=397&kat3=